CLINICAL TRIAL: NCT03120819
Title: A Randomized Controlled Trial to Determine the Effect of Supplementing an Oncologist's Recommendation to Exercise With Multimedia on Fatigue Levels in Breast Cancer Patients
Brief Title: Exercise Information for Women With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kerri Winters, Research Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00005997
Record Dates: First submitted 2017-04-12; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Cancer
Keywords: exercise; fatigue; physical activity
MeSH Terms: conditions — Neoplasms; Motor Activity; Fatigue

STUDY DESIGN:
Intervention Model Description: 2 x 3 repeated measures design with 2 groups and 3 time points
Who Masked: Care Provider, Investigator
Masking Description: Participant are randomized after receiving an exercise recommendation by their oncologist and thus oncologists are masked; however, study staff will administer survey questions including acceptability of the DVD and thus outcomes assessors are not masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oncologist Recommendation only (Active Comparator): Medical providers in this study provide a standardized brief recommendation for exercise to a consenting patient during a clinical visit. Patients randomized to this arm receive a packet that contained a study information sheet and standard published exercise information materials. The standard materials consisted of publicly available exercise recommendations for cancer survivors from the American Cancer Society (ACS). The packet of exercise information intended to represent general information about exercise and cancer that would be readily available to patients through the internet, a medical clinic, or cancer support services.
  Interventions: Behavioral: Oncologist Recommendation
- Oncologist Recommendation + DVD (Experimental): Participants in this arm receive the same oncologist's recommendation and written materials as the comparator group and also received an instructional yoga DVD. Inclusion of the video is intended to provide patients with a tool for following the oncologist's exercise recommendation. The instructional video contains a brief introduction from a breast cancer survivor, who was also featured in the exercise portion of the DVD, and safety information about lymphedema from a lymphedema therapist. The exercise program is a 30-minute, low intensity, restorative yoga program to improve whole body flexibility and to be safe for participants who were in active treatment for cancer and/or who had metastatic disease. Women are encouraged to use the DVD at least 3 times per week.
  Interventions: Behavioral: Oncologist Recommendation + DVD

INTERVENTIONS:
Behavioral: Oncologist Recommendation — Patients in this arm receive a 2-3 minute verbal recommendation about exercise from their treating oncologist
  Arms: Oncologist Recommendation only
Behavioral: Oncologist Recommendation + DVD — Patients in this arm receive a 2-3 minute verbal recommendation about exercise from their treating oncologist and then be sent an instructional exercise DVD to follow at their home three times per week for eight weeks
  Arms: Oncologist Recommendation + DVD

SUMMARY:
Fatigue is a troublesome symptom for breast cancer patients, which might be mitigated with exercise. Cancer patients often prefer their oncologist recommend an exercise program, yet a recommendation alone may not be enough to change behavior. Our study will determine whether adding an exercise DVD to an oncologist's recommendation to exercise led to better outcomes than a recommendation alone.

DETAILED DESCRIPTION:
Purpose: Controlled, intervention trials suggest that exercise may be a useful strategy to manage symptoms and side effects associated with cancer treatment. However, practical programs that facilitate exercise engagement among cancer patients are few and have been insufficiently studied. Medical providers may be best suited to deliver exercise information because of their frequent patient contact and the trust that patients place in their advice; however, unless sufficient resources are supplied in conjunction with verbal advice, patients may be less likely to successfully follow their physician's advice. The addition of an easy-to-follow, cancer specific exercise instructional video (DVD) to a provider's recommendation to exercise may provide patients with the motivation and ability to increase physical activity. We propose a feasibility study that will 1) determine acceptance and use of a provider-disseminated instructional home-exercise DVD among female cancer patients treated at OHSU and 2) determine if this cancer specific home-based DVD exercise program leads to greater decreases in fatigue, increases in exercise motivation and in physical activity compared to a standard exercise recommendation only among breast cancer patients treated at OHSU (N=100).

Methods: Medical providers who see female cancer patients during routine clinical visits will be approached to participate in the study. Willing providers will be enlisted to consent patients to receive a brief conversation (2-3 minutes) about the importance of exercise in their cancer care and then ask whether or not patients are willing to receive more information about the study from study staff. Providers will inform study staff about consenting participants who will then be randomized to one of two groups in the order that they enrolled. Study staff will then contact participants by phone to further explain the study and confirm eligibility then ask questions about their treatment, symptoms, and physical activity history. Based on their randomly assigned group, participants will receive either a control packet of standard exercise information based on guidelines from the American Cancer Society or standard exercise information plus a cancer specific home-based exercise DVD program. Fatigue, motivation for exercise, physical activity and use / acceptability of exercise information (+/- DVD) will be reassessed at 4 and 8 weeks following enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer
* Scheduled for a clinical appointment with a surgical, radiation or medical oncologist at Oregon Health & Science University (OHSU)
* Capable of answering survey questions by phone

Exclusion Criteria:

* Not medically cleared to participate in low-intensity exercise

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 95 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2011-07-31 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Patient-Reported Fatigue | baseline, 4 and 8 weeks
  Fatigue will be measured with the Brief Profile of Mood States Fatigue subscale

SECONDARY OUTCOMES:
Change in self-efficacy for exercise | baseline, 4 and 8 weeks
  Self-efficacy for exercise will be measured using the Self-Efficacy Assessment scale modified for exercise
Change in exercise readiness assessed by the Stage of Change for exercise | baseline, 4 and 8 weeks
  We will measure a person's readiness to engage in recommended levels of physical activity using the Stage of Change for behavior change modified for exercise
Change in self-report physical activity measured with the International Physical Activity Questionnaire | Baseline, 4 and 8 weeks
  We will measure changes in the reported time spent in physical activities per week

CONTACTS AND LOCATIONS:
Locations (1):
- OHSU School of Nursing, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Winters-Stone KM, Moe EL, Perry CK, Medysky M, Pommier R, Vetto J, Naik A. Enhancing an oncologist's recommendation to exercise to manage fatigue levels in breast cancer patients: a randomized controlled trial. Support Care Cancer. 2018 Mar;26(3):905-912. doi: 10.1007/s00520-017-3909-z. Epub 2017 Sep 30. PMID 28965138